CLINICAL TRIAL: NCT00458679
Title: Prolonged Immunization With Autologous CD40 Ligand and IL-2-Expressing Tumor Cells for Treatment of B-Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Treatment of B-Chronic Lymphocytic Leukemia (B-CLL) With Autologous CD40 Ligand and IL-2-Expressing Tumor Cells
Acronym: PRIMAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Professor/Director Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19747-PRIMAL; PRIMAL (Other: BCM IRB); NCT00602121 (obsolete NCT alias)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: CHRONIC LYMPHOCYTIC LEUKEMIA (B-CLL); CD40 LIGAND AND IL-2-EXPRESSING TUMOR CELLS
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — CD40 Ligand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): autologous B-CLL vaccine expressing CD40L and IL2
  Interventions: Biological: CD40 LIGAND AND IL-2-EXPRESSING TUMOR CELLS VACCINE

INTERVENTIONS:
Biological: CD40 LIGAND AND IL-2-EXPRESSING TUMOR CELLS VACCINE — Patients will receive a fixed dose (2 x 10^7) of IL-2 secreting B-cells together with (2 x 10^7)hCD40L expressing B-cells. They will receive 18 deltoid injections over 52 weeks.

SUMMARY:
We would like patients to be in a research study to determine the safety and effectiveness of special cells that may make their own immune system fight their cancer.

To do this, we will put a special gene into cancer cells that have been taken from the patients body. This will be done in the laboratory. This gene will make the cells produce interleukin 2 (IL-2), which is a natural substance that may help their immune system kill cancer cells. Additionally, we will stimulate the cancer cells with normal embryonic fibroblasts (cells that develop into normal connective tissues in the body) so that they will make another natural protein called CD40 ligand (CD40L). Studies of cancers in animals suggest IL-2 performs better when mixed with CD40L.

Some of these cells will then be put back into the patients body with the goal that they will act like a vaccine and stimulate their immune system to attack the CLL cells. Studies of cancers in animals and in cancer cells that are grown in laboratories suggest that combining substances like IL-2 and CD40L with cancer cells help the body recognize and kill cancer cells. We have already conducted a study similar to this in patients with CLL. In that study, the subjects received about three months of injections (shots). In those subjects we saw some changes in the subject's immune system that might indicate that the modified cells were helping their immune system fight the cancer. However, in most of the subjects this change in the immune system went away after the injections were stopped.

In this study we want to see if we can make the change in the immune system last longer by giving more injections over a longer period of time. We hope that this might produce a better response directed at the CLL cells. We will also be looking at the effect on cells called cancer stem cells which grow into the CLL cells we see in the blood. Specifically, this study will allow subjects to receive the injections for up to one year.

DETAILED DESCRIPTION:
Previously, some of the cancer cells taken from the patients body were separated in the laboratory and a specially produced human virus (adenovirus) that carries the IL-2 gene was put into the cells. Adenovirus is a common virus found in human respiratory systems. In its normal state, it can reproduce and cause a respiratory infection. Respiratory illnesses caused by adenovirus infections range from the common cold to pneumonia, croup and bronchitis. This adenovirus has been changed in the laboratory so that it is not likely to reproduce or cause an infection once it is in the patients body. The gene transfer method used in this study tries to add copies of the IL2 gene that increases the immune response against a tumor.

The rest of the cancer cells have been stimulated to express on their surface a substance called the human CD40L. These substances (IL-2 and CD40L), already naturally present in the patients body, are meant to help the immune system fight the cancer. In this study, the modified cancer cells will be injected under the skin. The patient will normally have the shots as an outpatient. The patient will receive the first eight (8) shots at 1-2 week intervals. They will then receive four (4) shots at 4 weekly intervals. After these first twelve shots, we will assess how the cancer is responding to these modified cells. If the cancer is not getting worse, the patient may receive an additional six (6) shots. These shots will again be given at 4 weekly intervals. In total, the patient may receive up to eighteen (18) shots over a period of one year. These shots must be given at the Methodist Hospital. Following these injections, the patient will be seen yearly for check-ups for 2 years after the first injection.

TESTS DURING AND AFTER EXPERIMENTAL TREATMENT:

A complete history and physical examination is necessary before the patient can be enrolled in the study. A physical examination will also be performed each time they are receive a shot of the modified cells. The place on the body where the patient has received their shots will be examined during the physical exam.

As mentioned above, the patient will then have yearly checkups for the 2 years after the first injection. After this, we will call the patients physician for updates on the patients health. These calls will be made annually until 5 years after the first injection.

To study how the modified cells are working in the body, we will take blood samples prior to each shot, then every four weeks for six months after the last injection, and then 2 years after the first injection.

The amount of blood that will be obtained for these tests is approximately 2-3 tablespoonfuls, which is considered to be a safe amount. If the patient has a central line (an IV line that has been placed in a large blood vessel that is meant to be used for long periods of time), the blood will be taken from it, so that extra "sticks" should not be needed. Additional office visits may be necessary to obtain this blood. The maximum total amount of blood to be collected from the patient is 78 tablespoons.

ELIGIBILITY:
INCLUSION CRITERIA:

Eligibility for blast collection:

* Patients are eligible for administration of their vaccine if they present with B-CLL (not in Richter's transformation) with measurable disease.
* Procurement consent signed and faxed to Research Coordinator
* Eligibility for Vaccine Administration (protocol entry)
* Manipulated B-CLL cells available (at least 12 injections)
* Patients are eligible for administration of their vaccine if they present with B-CLL (not in Richter's transformation) with measurable disease
* Patients must have a life expectancy of at least 10 weeks.
* Patients must have ECOG performance status of 0-2 as below:

  * Grade 0: Up and about, no restriction
  * Grade 1: Ambulatory, no strenuous activity
  * Grade 2: Ambulatory, capable of self-care appropriate for age. Up and about > 50% of time, but unable to carry out any physical activities or attend school.
  * Grade 3: Limited self-care only. Up and about < 50% of time
  * Grade 4: Disabled, no self-care. Bedridden or confined to chair
* Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study, and must have an absolute neutrophil count (ANC) of greater than or equal to 500/uL, absolute lymphocyte count (ALC) greater than or equal to 200/uL, hemoglobin greater than or equal to 8 g/dL and platelet count greater than or equal to 50,000/uL.
* Patients must be willing to practice appropriate birth control methods during the study and for 3 months after the study is concluded. This includes total abstinence, oral contraceptives, an intrauterine device, contraceptive implants under the skin, contraceptive injections (Depo-Provera [Registered]). Contraceptive foam with a condom is allowed. The male partner should use a condom.
* Patients must have adequate liver function (total bilirubin less than or equal to 1.5 mg/dl, SGOT less than or equal to 3 times normal, normal prothrombin time).
* Patients must have adequate renal function (creatinine less than 3 times normal for age or creatinine clearance greater than 80 mg/min/1.73m^2).
* Patients must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side-effects. Patients will be given a copy of the consent form.
* Patient must not have received treatment with other investigational agents within the last 4 weeks.

EXCLUSION CRITERIA:

* Infected at time of protocol entry, or receiving antibiotics (other than prophylactic trimethoprim sulfamethoxazole).
* HIV positive
* Pregnant or lactating
* Suffering from an autoimmune disease (including active graft-versus-host disease-GvHD, refractory immune thrombocytopenia-ITP or refractory autoimmune hemolytic anemia-AIHA)
* Receiving immunosuppressive drugs
* Patients without adequate cardiac function (congestive heart failure, significant arrhythmia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To measure adverse events of patients receiving prolonged immunization with an autologous B-CLL vaccine expressing CD40L and IL2 | 10 weeks

SECONDARY OUTCOMES:
Measurement of MHC-restricted or unrestricted anti-tumor immune responses | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MB, PhD, Principal Investigator — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (1):
- The Methodist Hospital, Houston, Texas, United States